CLINICAL TRIAL: NCT01880489
Title: Multicomponent Intervention to Reduce Sexual Risk and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, H. Jonathon Rendina, Assistant Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA034661 (NIH); R01DA034661 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: HIV; Sexually Transmitted Infections; Substance Use
Keywords: transgender women; sexual risk; substance use; HIV prevention; behavioral intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI + CBST Intervention (Experimental): Seven sessions of Motivational Interviewing and Cognitive Behavioral Skills Training
  Interventions: Behavioral: MI + CBST Intervention
- Wait List Control Condition (No Intervention)

INTERVENTIONS:
Behavioral: MI + CBST Intervention — The intervention focuses on exploring health goals, creating an action plan, learning about the impact stress, stigma, and substance use can have on health, improving personal growth and social support, and connecting with resources. The first two sessions will be primarily Motivational Interviewing and will explore participants' feelings about their sexual risk, substance use, non-medically monitored hormone and silicone use, and any other issues. Group sessions (Sessions 3-6) will incorporate Cognitive Behavioral Skills Training focusing barriers to physical and mental health. The last session will focus on reviewing progress toward health goals, identifying barriers to change, and generating a plan for connection to ongoing care to reach target health goals.
  Arms: MI + CBST Intervention

SUMMARY:
The objective is to expand and refine an intervention for transgender women (TW) into a 7-session individual- and group-based intervention that is scalable for community settings to reduce sexual risk and substance use and to increase stigma-coping and risk-buffering behaviors among TW in NYC. The investigators will pilot test the intervention with 20 TW and subsequently, conduct a randomized controlled trial with 240 TW to compare the intervention to a wait list control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Identify as a transgender woman (assigned male at birth and currently identify as female)
* Report 3 or more acts of unprotected anal or vaginal sex in the past 90 days and at least 1 in the past 30 days
* Report 5 or more days of illicit drug use in the past 90 days and at least 2 in the past 30
* Provide contact information
* Reside in the NYC metropolitan area
* Able to complete a survey in English (Spanish-language assistance can be provided by bilingual staff)
* Provide informed consent

Exclusion Criteria:

* Unstable, serious psychiatric symptoms
* Current suicidal/homicidal ideation
* Evidence of gross cognitive impairment
* Currently enrolled in a drug abuse treatment or enrolled in an HIV risk or drug use intervention study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Unprotected Sex Acts in the Past 90 Days | every 4 months over the course of 8 months
  Decreases from Baseline in the Number of Unprotected Sex Acts in the past 90 days at 4 and 8 months
Number of Days of Drug Use in the Past 90 Days | every 4 months over the course of 8 months
  Decreases from Baseline in the Number of Days of Drug Use in the past 90 days at 4 and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: H. Jonathon Rendina, Ph.D., Principal Investigator — Hunter College of City University of New York
Locations (1):
- Center for HIV/AIDS Educational Studies and Training of Hunter College, CUNY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No